CLINICAL TRIAL: NCT04323553
Title: Comparison of Pulsed-field Gel Electrophoresis and Whole Genome Sequencing to Determine Transmission Rate of ESBL-producing E.Coli
Acronym: PFGE-WGS
Status: Terminated | Type: Observational
Why Stopped: This study is no longer of interested as one of the technology used is already outdated.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00188
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Analysis Transmission Rate
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Enterobacteriaceae
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESBL E.coli strains from 24 contact-index patients: 48 ESBL-E. coli strains from 24 contact-index patients
  Interventions: Diagnostic Test: Pulsed-field gel electrophoresis and whole genome sequencing; Other: Data collection

INTERVENTIONS:
Diagnostic Test: Pulsed-field gel electrophoresis and whole genome sequencing — Comparison of the two different techniques
Other: Data collection — Demographic data (age, gender, hospital admission and discharge date, rooms and wards with dates of admission and discharge, hospitalization prior to current hospital stay, discharge destination, outcome, cause of death, travel history, recent hospitalization in an ESBL-high burden region, admission from another healthcare facility, admission from a long-term care facility, occupational or household contact to animals) Clinical data (date of diagnosis of ESBL-producing E. coli carriage, type of infection/colonization with ESBL- producing E. coli, comorbidities, Charlson Comorbidity Index, infectious diseases after detection of ESBL-PE, active open wounds, indwelling vascular devices, urinary catheterization) Treatment data (Immunosuppression, antibiotic therapy, concomitant medication and surgical therapy prior to and during hospital stay) Microbiological data

SUMMARY:
The aim of this quality control study is to compare two different techniques to determine ESBL-producing E.coli transmission.

DETAILED DESCRIPTION:
Pulse-field gel electrophoresis (PFGE) was considered the reference standard to determine transmission events of extended-spectrum Beta-Lactamase (ESBL) producing E.coli . However, this technique lacks the resolution to differentiate closely related strains, which is needed to identify ESBL-transmission. Furthermore, PFGE is not able to distinguish mobile genetic elements. In contrast, whole genome sequencing (WGS) allows the identification of single-nucleotide polymorphisms (SNPs) that differentiate bacterial strains and mobile genetic elements, such as plasmids at the highest possible resolution, therefore enabling investigation of their relatedness by phylogenetic analyses and ultimately detailed exploration of transmission pathways. As WGS is now readily available and affordable, the investigators aim to reinvestigate transmission events in the 24 index-contact patient-pairs identified after cessation of contact precautions by reassessing the genetic relatedness of both strains and mobile genetic elements by sequencing all 48 recovered ESBL- E.coli strains.

The investigators hypothesize that the number of transmission events as defined by transmission of ESBL-producing E. coli strains may have been overestimated by PFGE as compared to WGS, as PFGE lacks the resolution to differentiate closely related strains. However, transmission of mobile genetic elements may have been missed by PFGE as this technology is not able to identify the genetic relatedness of plasmids, genes and other mobile genetic elements. Thus WGS may reveal additional transmission events defined as the transmission of mobile genetic elements.

Different sequencing approaches may yield different results in terms of detection of transmission events.

The investigators hypothesize that short-read sequencing may suffice to reliably detect relatedness of strains but that additional long-read sequencing approaches are needed to detect transmission of mobile genetic elements.

ELIGIBILITY:
Inclusion Criteria:

* The patient population is defined as the 24 contact-index patient pairs identified during screening of contact patients after cessation of contact precautions as part of a quality control, performed from June 2012 to December 2013 at the University Hospital Basel and from January 2012 to December 2013 at the FELIX PLATTER-Hospital.

Exclusion Criteria:

* Patients not meeting the above mentioned inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population is defined as the 24 contact-index patient pairs identified during screening of contact patients after cessation of contact precautions during June 2012 to December 2013 at the University Hospital Basel and from January 2012 to December 2013 at the FELIX PLATTER-Hospital.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Number of transmission events as determined by WGS | January 2012- December 2020
  Transmission events will be categorized into transmission of strains and transmission of mobile genetic elements. The number of transmission events as determined by WGS will be compared to the number of transmission events as determined by PFGE. Patient-related characteristics and exposures will be compared between patients with and without transmission events.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin Sutter, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland